CLINICAL TRIAL: NCT05443308
Title: Cerebral Vascular Reserve in Small Vessel Disease and Alzheimers Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lisbeth Marner, MD, Associate professor, Bispebjerg Hospital
Other Study IDs: H-21076058
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease; Dementia, Vascular
Keywords: Positron-Emission Tomography; Perfusion
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer Disease: patients with presumed Alzheimer disease and no known vascular, psychiatric or other major diseases age > 60 years
  Interventions: Diagnostic Test: Cerebral [15O]H2O PET before and after diamox infusion
- Small vessel disease: patients diagnosed with small vessel disease of the brain by MRI and presumed cognitive dysfunction and no other known psychiatric or other major diseases.
  age > 60 years
  Interventions: Diagnostic Test: Cerebral [15O]H2O PET before and after diamox infusion
- Healthy subjects: Age-matched subjects with no known vascular, psychiatric or other major diseases.
  age > 60 years
  Interventions: Diagnostic Test: Cerebral [15O]H2O PET before and after diamox infusion

INTERVENTIONS:
Diagnostic Test: Cerebral [15O]H2O PET before and after diamox infusion — Cerebral [15O]H2O PET before and after diamox infusion

SUMMARY:
Alzheimers disease and cerebral small vessel disease have a considerably overlap in patients and have common risk factors. The diseases are difficult to separate in individual patients and we hypothesize that a reduced cerebral vascular reserve may be a measurement of small vessel disease independent of Alzheimers disease.

Patients with presumed Alzheimers disease (n=20), cerebral small vessel disease (n=20) and healthy age-matched subjects (n=15) are examined with quantitative [15O]H2O positron emission tomography (PET) for measurements of brain perfusion before and after diamox infusion that dilates cerebral vessels. Additional [15O]H2O PET scans of the heart allows for a non-invasive input function so the cerebral vascular reserve can be measured quantitatively.

DETAILED DESCRIPTION:
Alzheimers disease and cerebral small vessel disease are increasingly common in the elderly population and constitute around 90% of new dementia cases in Denmark. The diseases have a considerably overlap in patients and have common risk factors. The cause of dementia can be difficult to separate in individual patients but a reduced cerebral vascular reserve may be a measurement of small vessel disease independent of Alzheimers disease. We hypothesized that patient with small vessel disease have reduced increase in brain perfusion after medical brain vessel dilatation. While Alzheimer patients may have reduced perfusion in rest but normal increase after medical brain vessel dilatation as compared to healthy subjects.

Patients with presumed Alzheimers disease (n=20), cerebral small vessel disease (n=20) and healthy age-matched subjects (n=15) are examined with quantitative [15O]H2O PET for measurements of brain perfusion before and after diamox infusion that dilates cerebral vessels. Additional [15O]H2O PET scans of the heart allows for a non-invasive input function so the cerebral vascular reserve can be measured quantitatively.

ELIGIBILITY:
Inclusion Criteria:

* presumed Alzheimer's Disease (group 1)
* diagnosed with small vessel disease of the brain by MRI and presumed cognitive dysfunction (group 2)

Exclusion Criteria:

* major claustrophobia
* major psychiatric diseases
* other major somatic diseases
* allergy to diamox

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited from Department of Neurology, and Department of Geriatric and Palliative Medicine at Bispebjerg Hospital, Copenhagen, Denmark.
  Healthy subjects are recruited from internet advertisments.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Vascular reserve perfusion | 20 min after diamox infusion
  Brain perfusion after diamox infusion (mL / min / 100 g tissue)
Vascular reserve change | 20 min after diamox infusion
  Change in Brain perfusion after diamox infusion (mL / min / 100 g tissue and %) compared to before diamox infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine, Copenhagen University Hospital Bispebjerg, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available at reasonable request following Danish laws on personal data regulations.